CLINICAL TRIAL: NCT01079234
Title: A 26-week Trial Investigating the Dosing Flexibility, Efficacy and Safety of NN1250 in Subjects With Type 1 Diabetes With a 26-week Extension (Begin™: Flex T1)
Brief Title: Comparison of NN1250 With Insulin Glargine in Type 1 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3770; U1111-1112-8813 (Other: WHO); 2009-012923-27 (EudraCT Number)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flex + insulin aspart (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- Fixed + insulin aspart (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IGlar + insulin aspart (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily
  Arms: Fixed + insulin aspart; Flex + insulin aspart
Drug: insulin glargine — Insulin glargine injected subcutaneously (under the skin) once daily
  Arms: IGlar + insulin aspart
Drug: insulin aspart — At least three daily doses at meal-time

SUMMARY:
This trial is conducted in Europe and in the United States of America (USA). The aim of this trial is to investigate the efficacy and safety of NN1250 (insulin degludec) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for 12 months or longer, hereof the last 3 months with injection based therapies
* Current treatment with any basal insulin (e.g. insulin glargine, insulin detemir, NPH insulin) using one or two daily injections and with three or more daily meal-time insulin injections (e.g. insulin aspart, insulin lispro, insulin glulisine, human insulin) used as bolus insulin therapy
* HbA1c maximum 10.0 % by central laboratory analysis
* Body Mass Index (BMI) below or equal to 35.0 kg/m^2
* Ability to self-manage insulin therapy as assessed by confirmation (verbal confirmation at screening visit) of a changed insulin dose in the preceding two months prior to screening
* Ability and willingness to adhere to the protocol including performance of self measured plasma glucose (SMPG) profiles and self adjustment of insulin doses

Exclusion Criteria:

* Use within the last 3 months prior to Visit 1 of any antidiabetic glucose lowering drug other than insulin
* Cardiovascular disease, within the last 6 months prior to visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/ untreated severe hypertension (systolic blood pressure above or equal to 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure above or equal to 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (74):
- United States (37):
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Redondo Beach, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, DeLand, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Nampa, Idaho
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Springfield, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Flemington, New Jersey
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Spokane, Washington
- Belgium (5):
  - Novo Nordisk Investigational Site, Aalst
  - Novo Nordisk Investigational Site, Arlon
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Leuven
- Germany (8):
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Rehburg-Loccum
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Völklingen
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Norway (6):
  - Novo Nordisk Investigational Site, Ålesund
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Stavanger
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Warsaw
- United Kingdom (12):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Inverness
  - Novo Nordisk Investigational Site, Ipswich
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Southall
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Welwyn Garden City

REFERENCES:
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Heller S, Mathieu C, Kapur R, Wolden ML, Zinman B. A meta-analysis of rate ratios for nocturnal confirmed hypoglycaemia with insulin degludec vs. insulin glargine using different definitions for hypoglycaemia. Diabet Med. 2016 Apr;33(4):478-87. doi: 10.1111/dme.13002. Epub 2015 Dec 13. PMID 26484727
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Seufert J, Solberg H, Kinduryte O, Johansen T, Hollander P. Insulin degludec does not increase antibody formation versus insulin glargine: an evaluation of phase IIIa trials. Diabetes Obes Metab. 2016 Jul;18(7):716-20. doi: 10.1111/dom.12621. Epub 2016 Feb 8. PMID 26663320
- [Derived] Mathieu C, Hollander P, Miranda-Palma B, Cooper J, Franek E, Russell-Jones D, Larsen J, Tamer SC, Bain SC; NN1250-3770 (BEGIN: Flex T1) Trial Investigators. Efficacy and safety of insulin degludec in a flexible dosing regimen vs insulin glargine in patients with type 1 diabetes (BEGIN: Flex T1): a 26-week randomized, treat-to-target trial with a 26-week extension. J Clin Endocrinol Metab. 2013 Mar;98(3):1154-62. doi: 10.1210/jc.2012-3249. Epub 2013 Feb 7. PMID 23393185
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main/extension trial periods were conducted at 71/68 sites in 6 countries:
  Belgium (5/5 sites), Germany (7/7 sites), Norway (5/5 sites), Poland (5/5 sites), United Kingdom (UK) (12/11 sites), and United States of America (U.S.) (37/35 sites). 57 patients did not participate in the extension trial.
Pre-assignment Details: All subjects who completed the 26-week main trial and were found to be eligible for the extension trial were offered to participate in the 26-week extension trial (NCT01079234). Total duration of trial was up to 52 weeks (26 weeks+ 26 weeks) with two times 7-12 day follow-up periods.
Groups:
- IDeg OD FF: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (s.c.) with alternating morning and evening dosing according to a fixed flexible (FF) schedule (approximately 8-40 hours intervals) in combination with insulin aspart (IAsp) for 26 weeks in main period. Insulin doses were individually adjusted by the subjects.
- IDeg OD: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (s.c.) with the evening meal in combination with insulin aspart (IAsp) for 26 weeks in main period. Insulin doses were individually adjusted by the subjects.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) subcutaneously (s.c.) according to local labelling in combination with insulin aspart (IAsp) for 52 weeks (26 weeks in main period + 26 weeks in extension period). Insulin doses were individually adjusted by the subjects.
- IDeg OD F: The subjects randomised to the 2 insulin degludec (IDeg) treatment arms in the main period (IDeg OD FF and IDeg OD) were pooled into this IDeg OD Free Flex arm (IDeg OD F). IDeg was given once daily (OD) subcutaneously (s.c.) at any time of the day (approximately 8-40 hours intervals) in combination with insulin aspart (IAsp) for 26 weeks in the extension period (52 weeks in total). Insulin doses were individually adjusted by the subjects.
Period: Main: Week 0 to 26
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD | IDeg OD F
Started | 164 | 165 | 164 | 0
Exposed | 164 | 165 | 161 (Three subjects withdrew prior to exposure to trial drug.) | 0
Completed | 138 | 139 | 152 | 0
Not Completed | 26 | 26 | 12 | 0
Not completed — Adverse Event | 5 | 4 | 1 | 0
Not completed — Lack of Efficacy | 2 | 1 | 1 | 0
Not completed — Protocol Violation | 6 | 2 | 4 | 0
Not completed — Withdrawal criteria | 6 | 6 | 2 | 0
Not completed — Unclassified | 7 | 13 | 4 | 0
Period: Extension: Week 27 to 52
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD | IDeg OD F
Started | 0 | 0 | 133 (Nineteen subjects from main trial did not continue into extension trial) | 239 (Thirty eight subjects did not continue into extension trial.)
Completed | 0 | 0 | 122 | 223
Not Completed | 0 | 0 | 11 | 16
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 2 | 5
Not completed — Withdrawal criteria | 0 | 0 | 4 | 2
Not completed — Unclassified | 0 | 0 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 164 | 165 | 164 | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.4) | 44.5 (13.1) | 44.1 (12.6) | 43.7 (13.1)
Gender [Count of Participants; unit: Participants]
  Female | 62 | 71 | 76 | 209
  Male | 102 | 94 | 88 | 284
HbA1c (glycosylated haemoglobin) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.7 (1.0) | 7.7 (0.9) | 7.7 (0.9) | 7.7 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.6 (4.1) | 10.0 (4.0) | 9.7 (4.2) | 9.8 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 26 Weeks of Treatment
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Number analyzed (Participants) | 164 | 165 | 164
percentage of glycosylated haemoglobin | -0.40 (0.59) | -0.41 (0.71) | -0.58 (0.72)

2. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment.
Time Frame: Week 0, Week 52
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). The subjects randomised to 2 IDeg arms during the main trial were pooled into the IDeg OD F in extension trial.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IGlar OD | IDeg OD F
Number analyzed (Participants) | 164 | 329
percentage of glycosylated haemoglobin | -0.21 (0.73) | -0.13 (0.67)

3. Secondary Outcome: Main Trial (Secondary Endpoint): Change in Fasting Plasma Glucose (FPG) After 26 Weeks of Treatment
Description: Change from baseline in FPG after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). For 6 subjects baseline values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Number analyzed (Participants) | 161 | 164 | 162
mmol/L | -1.28 (5.03) | -2.54 (5.11) | -1.33 (5.21)

4. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Fasting Plasma Glucose (FPG) After 52 Weeks of Treatment
Description: Change from baseline in FPG after 52 weeks of treatment.
Time Frame: Week 0, Week 52
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). FPG baseline values were missing for 6 subjects. The subjects randomised to 2 IDeg arms during the main trial were pooled into the IDeg OD F in extension trial.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IGlar OD | IDeg OD F
Number analyzed (Participants) | 162 | 325
mmol/L | -0.61 (5.23) | -1.73 (5.32)

5. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator. The subjects randomised to 2 IDeg arms during the main trial were pooled into the IDeg OD F in extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IGlar OD | IDeg OD F
Number analyzed (Participants) | 161 | 329
Episodes/100 years of patient exposure | 6341 | 6811

6. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.The subjects randomised to 2 IDeg arms during the main trial were pooled into the IDeg OD F in extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IGlar OD | IDeg OD F
Number analyzed (Participants) | 161 | 329
Episodes/100 years of patient exposure | 848 | 640

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 52 weeks + 7 days follow up
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg OD F | IGlar OD
Serious Adverse Events (participants affected / at risk) | 25/329 | 12/161
Other Adverse Events (participants affected / at risk) | 187/329 | 105/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD F (N=329) | IGlar OD (N=161)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (12) | 4 (4)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 2 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudo aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyper osmolar state (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD F (N=329) | IGlar OD (N=161)
Diarrhoea (Gastrointestinal disorders) | 9 (15) | 12 (15)
Nausea (Gastrointestinal disorders) | 18 (21) | 8 (13)
Vomiting (Gastrointestinal disorders) | 18 (22) | 11 (12)
Gastroenteritis (Infections and infestations) | 19 (22) | 6 (6)
Nasopharyngitis (Infections and infestations) | 99 (174) | 48 (85)
Sinusitis (Infections and infestations) | 23 (28) | 13 (18)
Upper respiratory tract infection (Infections and infestations) | 28 (39) | 21 (30)
Wrong drug administered (Injury, poisoning and procedural complications) | 18 (19) | 7 (8)
Hypoglycaemia (Metabolism and nutrition disorders) | 24 (38) | 13 (42)
Headache (Nervous system disorders) | 33 (61) | 24 (48)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 11 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (36) | 14 (15)
Gastroenteritis viral (Infections and infestations) | 9 (11) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.